CLINICAL TRIAL: NCT02795052
Title: Neurologic Bone Marrow Derived Stem Cell Treatment Study
Brief Title: Neurologic Stem Cell Treatment Study
Acronym: NEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MD Stem Cells (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDSC-NEST
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-04

CONDITIONS: Neurologic Disorders; Nervous System Diseases; Neurodegenerative Diseases; Neurological Disorders; Stroke; Traumatic Brain Injury; Cadasil; Chronic Traumatic Encephalopathy; Cerebral Infarction; Cerebral Ischemia; Cerebral Stroke; Cerebral Hemorrhage; Parkinson; Multi-System Degeneration; MSA - Multiple System Atrophy; Progressive Supranuclear Palsy; ALS; Amyotrophic Lateral Sclerosis; Neuropathy; Diabetic Neuropathies; Alzheimer Disease; Dementia; Frontotemporal Dementia; Lewy Body Disease; Cognitive Impairment; Lewy Body Variant of Alzheimer Disease
Keywords: Neurologic Disease; Cerebral Vascular Accident; Stroke; Traumatic Brain Injury; Multiple Sclerosis; Parkinsons Disease; Neuropathy; Diabetic Neuropathy; Cerebral Ischemia; Cognitive Impairment; Dementia; Neurodegeneration
MeSH Terms: conditions — Nervous System Diseases; Neurodegenerative Diseases; Stroke; Brain Injuries, Traumatic; CADASIL; Chronic Traumatic Encephalopathy; Cerebral Infarction; Brain Ischemia; Cerebral Hemorrhage; Shy-Drager Syndrome; Supranuclear Palsy, Progressive; Amyotrophic Lateral Sclerosis; Diabetic Neuropathies; Alzheimer Disease; Dementia; Frontotemporal Dementia; Lewy Body Disease; Cognitive Dysfunction; Lewy Body Variant of Alzheimer Disease; Multiple Sclerosis; Parkinson Disease; Nerve Degeneration

STUDY DESIGN:
Intervention Model Description: Intravenous and intranasal bone marrow derived stem cells.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1- Intravenous and Intranasal BMSC (Other): Intervention- Autologous bone marrow aspiration and separation of Bone Marrow Derived Stem Cell (BMSC) fraction then provided intravenously and intranasally (lower 1/3 of nasal passages).
  Interventions: Procedure: Intravenous and Intranasal BMSC

INTERVENTIONS:
Procedure: Intravenous and Intranasal BMSC — Autologous Bone Marrow Derived Stem Cells provided intravenous and intranasal (lower 1/3 of nose)
  Other Names: IV and IN BMSC

SUMMARY:
This is a human clinical study involving the isolation of autologous bone marrow derived stem cells (BMSC) and transfer to the vascular system and inferior 1/3 of the nasal passages in order to determine if such a treatment will provide improvement in neurologic function for patients with certain neurologic conditions. http://mdstemcells.com/nest/

DETAILED DESCRIPTION:
Various clinical studies have registered with the National Institutes of Health (NIH) to study neurologic diseases and damage. There have also been a number of journal reports of the benefits of treatment with BMSC for diseases and damage to nervous tissue. The investigators hope to add to the volume of literature regarding the use of BMSC in those neurologic diseases and conditions identified as likely to respond to this treatment.

Intravenous administration of BMSC is a well-established approach to neurologic disease and injury with much support for its effectiveness in the pre-clinical and clinical literature. BMSC and the associated bone marrow fraction are posited to have a number of different mechanisms by which they may potentially improve neurologic function. In regards their ability to penetrate the blood-brain barrier for potential neuronal transdifferentiation and direct impact on the neurons and glial tissue within the brain, it should be remembered that within the diencephalon there are specific circumventricular organs which lie in the wall of the third ventricle. These are noteworthy for a significantly diminished blood-brain barrier and glial limitans which facilitates their function of coordinating homeostatic mechanisms of the endocrine and nervous systems. Therefore the investigators believe entry of BMSC may be facilitated in this area of the brain.

The NEST Study provides a treatment Arm 1 which combines intravenous BMSC with topical application of BMSC to the lower 1/3 of the nasal passages as a means of introducing BMSC to the Central Nervous System (CNS). This is applied bilaterally to the inferior nasal conchas and meatuses. The Trigeminal Nerve or 5th Cranial Nerve is a paired, large sensory and motor nerve with multiple branches. It provides sensation to the surface and interior structures of the face including the nasal mucosa that lines the nose. The nerves of the Trigeminal Nerve providing sensation to this area converge and enter the brain at the level of the pons. There is documentation in the scientific literature that intranasal delivery of BMSC allows the BMSC to follow the pathways of the trigeminal nerve, facilitating entry into the parenchyma and cerebral spinal fluid (CSF) for effects on the CNS.

ELIGIBILITY:
Inclusion Criteria:

1. Have documented functional damage to the central or peripheral nervous system unlikely to improve with present standard of care.
2. Be at least 6 months post-onset of the disease.
3. If under current medical therapy (pharmacologic or surgical treatment) for the condition be considered stable on that treatment and unlikely to have reversal of the associated neurologic functional damage as a result of the ongoing pharmacologic or surgical treatment.
4. In the estimation of Dr. Weiss and the neurologists have the potential for improvement with BMSC treatment and be at minimal risk of any potential harm from the procedure.
5. Be over the age of 18 and capable of providing informed consent.
6. Be medically stable and able to be medically cleared by their primary care physician or a licensed primary care practitioner for the procedure. Medical clearance means that in the estimation of the primary care practitioner, the patient can reasonably be expected to undergo the procedure without significant medical risk to health.

Exclusion Criteria:

1. All patients must be capable of an adequate neurologic examination and evaluation to document the pathology. This will include the ability to cooperate with the exam.
2. Patients must be capable and willing to undergo follow up neurologic exams with the sub-investigators or their own neurologists as outlined in the protocol.
3. Patients must be capable of providing informed consent.
4. In the estimation of Dr. Weiss the BMSC collection and treatment will not present a significant risk of harm to the patient's general health or to their neurologic function. .
5. Patients who are not medically stable or who may be at significant risk to their health undergoing the procedure will not be eligible.
6. Women of childbearing age must not be pregnant at the time of treatment and should refrain from becoming pregnant for 3 months post treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Neurologic Function | 0,1,3,6 and 12 months
  Neurologic function from prior to treatment (0 month) and the change in neurologic function at 1,3,6 and 12 months post treatment will be compared to pretreatment using the Neuro-QOL (Neurology Quality of Life) questionnaire. The scales of the Neuro-QOL assess the following Outcome Measures: Communication, Social Roles and Activities ,Anxiety , Depression, Emotional and Behavioral Dyscontrol, Lower Extremity Function (Mobility), Positive Affect and Well-Being, Sleep Disturbance, Upper Extremity Function ( Fine Motor, ADL/Activities of Daily Living) , Stigma , Satisfaction with Social roles and Activities, Cognitive Function. The scale for each question ranges from 1 to 5 with 1 being the most impairment and 5 being no impairment; higher numbers are better. The scale can range from 5 indicating no impairment to 45 for significant impairment. Each scale will be recorded and presented as separate Outcome Measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Levy, MD, Study Chair — MD Stem Cells; Jeffrey Weiss, MD, Principal Investigator — Coral Springs, Florida
Locations (3):
- United States (2):
  - MD Stem Cells, Westport, Connecticut
  - MD Stem Cells, Coral Springs, Florida
- The Saudi-German Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chapman CD, Frey WH 2nd, Craft S, Danielyan L, Hallschmid M, Schioth HB, Benedict C. Intranasal treatment of central nervous system dysfunction in humans. Pharm Res. 2013 Oct;30(10):2475-84. doi: 10.1007/s11095-012-0915-1. Epub 2012 Nov 8. PMID 23135822
- [Background] Jiang Y, Zhu J, Xu G, Liu X. Intranasal delivery of stem cells to the brain. Expert Opin Drug Deliv. 2011 May;8(5):623-32. doi: 10.1517/17425247.2011.566267. Epub 2011 Mar 19. PMID 21417782
- [Background] Bhasin A, Srivastava M, Bhatia R, Mohanty S, Kumaran S, Bose S. Autologous intravenous mononuclear stem cell therapy in chronic ischemic stroke. J Stem Cells Regen Med. 2012 Nov 26;8(3):181-9. doi: 10.46582/jsrm.0803011. eCollection 2012. PMID 24693196
- [Background] Teixeira FG, Carvalho MM, Sousa N, Salgado AJ. Mesenchymal stem cells secretome: a new paradigm for central nervous system regeneration? Cell Mol Life Sci. 2013 Oct;70(20):3871-82. doi: 10.1007/s00018-013-1290-8. Epub 2013 Mar 1. PMID 23456256
- [Background] Lescaudron L, Naveilhan P, Neveu I. The use of stem cells in regenerative medicine for Parkinson's and Huntington's Diseases. Curr Med Chem. 2012;19(35):6018-35. PMID 22963567
- [Background] Laroni A, de Rosbo NK, Uccelli A. Mesenchymal stem cells for the treatment of neurological diseases: Immunoregulation beyond neuroprotection. Immunol Lett. 2015 Dec;168(2):183-90. doi: 10.1016/j.imlet.2015.08.007. Epub 2015 Aug 18. PMID 26296458
- [Background] Anbari F, Khalili MA, Bahrami AR, Khoradmehr A, Sadeghian F, Fesahat F, Nabi A. Intravenous transplantation of bone marrow mesenchymal stem cells promotes neural regeneration after traumatic brain injury. Neural Regen Res. 2014 May 1;9(9):919-23. doi: 10.4103/1673-5374.133133. PMID 25206912
- [Background] Weiss JN, Levy S. Neurologic Stem Cell Treatment Study (NEST) using bone marrow derived stem cells for the treatment of neurological disorders and injuries: study protocol for a nonrandomized efficacy trial. Clin Trials Degener Dis. 2016 [cited 2019 Jun 18];1:176-80.
- [Background] Cella D, Lai JS, Nowinski CJ, Victorson D, Peterman A, Miller D, Bethoux F, Heinemann A, Rubin S, Cavazos JE, Reder AT, Sufit R, Simuni T, Holmes GL, Siderowf A, Wojna V, Bode R, McKinney N, Podrabsky T, Wortman K, Choi S, Gershon R, Rothrock N, Moy C. Neuro-QOL: brief measures of health-related quality of life for clinical research in neurology. Neurology. 2012 Jun 5;78(23):1860-7. doi: 10.1212/WNL.0b013e318258f744. Epub 2012 May 9. PMID 22573626
- [Background] Cella D, Nowinski C, Peterman A, Victorson D, Miller D, Lai JS, Moy C. The neurology quality-of-life measurement initiative. Arch Phys Med Rehabil. 2011 Oct;92(10 Suppl):S28-36. doi: 10.1016/j.apmr.2011.01.025. PMID 21958920